CLINICAL TRIAL: NCT01636960
Title: An Open-Label, Single-arm, Multicenter Phase I Study of SCH 54031 (Pegylated Interferon Alfa-2b) as an Adjuvant Treatment in Japanese Patients With Malignant Melanoma (Protocol No. MK-4031 370 Also Known as SCH 54031, P08556)
Brief Title: A Study of Pegylated Interferon Alfa-2b (MK-4031) as an Adjuvant Treatment in Japanese Patients With Malignant Melanoma (MK-4031-370)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated after 118 weeks from the study start, during the maintenance phase, due to regulatory approval in Japan.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08556; MK-4031-370 (Other: Merck protocol number); 132228 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants receiving PegIFN alfa-2b (Experimental): Participants receive PegIFN alfa-2b 6 µg/kg subcutaneously (SC) on Day 1 of each week for 8 weeks (Induction) and then 3 µg/kg SC once weekly for up to 252 weeks (Maintenance).
  Interventions: Biological: PegIFN alfa-2b

INTERVENTIONS:
Biological: PegIFN alfa-2b

SUMMARY:
This is a study to evaluate the safety and tolerability of peginterferon alfa-2b (PegIFN alfa-2b) as adjuvant treatment in Japanese participants with malignant melanoma after definitive surgical resection including complete lymphadenectomy. Participants on this study will initially receive PegIFN alfa-2b for 8 weeks (Induction Phase) and then may continue to receive PegIFN alfa-2b (Maintenance Phase) as long as they are experiencing clinical benefit (Up to 252 weeks). The primary hypothesis is that peginterferon alfa-2b administered on a weekly basis is safe and tolerated.

DETAILED DESCRIPTION:
The study was terminated after 118 weeks from the study start, during the maintenance phase, due to regulatory approval in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III melanoma
* Primary melanoma completely excised
* Full lymphadenectomy within 84 days prior to initiation of study treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Ocular melanoma or melanoma of the mucous membranes
* Evidence of distant or non-regional lymph node metastases
* In-transit melanoma
* Previously treated with interferon alpha/beta, chemotherapy, hormonal therapy, radiotherapy or immunotherapy/vaccine for melanoma

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12-25 (Actual); Primary Completion 2014-03-26 (Actual); Study Completion 2015-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yamazaki N, Uhara H, Wada H, Matsuda K, Yamamoto K, Shimamoto T, Kiyohara Y. Phase I study of pegylated interferon-alpha-2b as an adjuvant therapy in Japanese patients with malignant melanoma. J Dermatol. 2016 Oct;43(10):1146-1153. doi: 10.1111/1346-8138.13338. PMID 27087489
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P08556&kw=P08556&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled Japanese participants with Stage II or III malignant melanoma who had undergone surgical resection and lymphadenectomy.
Groups:
- Participants Receiving PegIFN Alfa-2b: Participants received PegIFN alfa-2b 6 µg/kg subcutaneously (SC) on Day 1 of each week for 8 weeks (Induction) and then 3 µg/kg SC once weekly for up to 252 weeks (Maintenance).
Period: Induction Phase
Arm/Group | Participants Receiving PegIFN Alfa-2b
Started | 9
Completed | 7 (Participants continuing into Maintenance Phase)
Not Completed | 2
Not completed — Adverse Event | 2
Period: Maintenance Phase
Arm/Group | Participants Receiving PegIFN Alfa-2b
Started | 7
Completed | 0
Not Completed | 7
Not completed — Continued drug after regulatory approval | 3
Not completed — Adverse Event | 3
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Receiving PegIFN Alfa-2b
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) - Induction Phase
Description: A DLT was an event (clinical or laboratory) that resulted in a change in the given dose.
Time Frame: From first dose to end of induction phase; up to 8 Weeks
Population: All participants in the induction phase of the study
Measure: Number; unit: Participants
Arm/Group | Participants Receiving PegIFN Alfa-2b
Number analyzed (Participants) | 9
Participants | 2

2. Secondary Outcome: Safety: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event was any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: From first dose through follow-up; up to 265 Weeks
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving PegIFN Alfa-2b
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Number of Participants Discontinuing Study Drug Because of AEs
Description: as for outcome 2
Time Frame: From first dose to last dose of treatment; up to 260 Weeks
Population: All participants receiving at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving PegIFN Alfa-2b
Number analyzed (Participants) | 9
Participants | 5

ADVERSE EVENTS:
Time Frame: From first dose through follow-up; up to 265 Weeks
Arm/Group | Participants Receiving PegIFN Alfa-2b
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving PegIFN Alfa-2b (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (5)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (3)
Eye pain (Eye disorders) | 1 (3)
Photophobia (Eye disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 2 (2)
Retinopathy (Eye disorders) | 2 (2)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (12)
Periodontal disease (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 6 (13)
Fatigue (General disorders) | 5 (7)
Injection site erythema (General disorders) | 3 (3)
Injection site extravasation (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 3 (3)
Injection site reaction (General disorders) | 6 (29)
Malaise (General disorders) | 6 (23)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 9 (33)
Adenoiditis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (2)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Pericoronitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (8)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 8 (11)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (6)
Neutrophil count decreased (Investigations) | 9 (21)
Platelet count decreased (Investigations) | 5 (7)
Weight decreased (Investigations) | 5 (6)
White blood cell count decreased (Investigations) | 9 (19)
Decreased appetite (Metabolism and nutrition disorders) | 4 (9)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (20)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (10)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 5 (63)
Insomnia (Psychiatric disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (3)
Ocular discomfort (Eye disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Injection site joint pain (General disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Quadriplegia (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated after 118 weeks from the study start, during the maintenance phase, due to regulatory approval in Japan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the trial without prior written consent of the Sponsor. The Investigator further agrees to provide review copies of abstracts or manuscripts (both oral and textual including transmission through any electronic medium). No publication or manuscript shall contain any trade secret information of the Sponsor or any proprietary or confidential information of the Sponsor.